CLINICAL TRIAL: NCT05126966
Title: A Phase IIIb, Multicenter, Randomized, Visual Assessor-Masked Study Of The Effectiveness And Safety Of A 36-Week Refill Regimen For The Port Delivery System With Ranibizumab Vs Aflibercept Treat & Extend In Subjects With Neovascular Age-Related Macular Degeneration
Brief Title: A Study Of The Effectiveness And Safety Of A 36-Week Refill Regimen For The Port Delivery System With Ranibizumab Vs Aflibercept Treat & Extend In Subjects With Neovascular Age-Related Macular Degeneration
Acronym: Diagrid
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Roche/Genentech has initiated an immediate pause of all new PDS implantations because the implants from commercial supply in the clinical studies did not meet the filed specifications for the intended use
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MR42410; 2021-003226-71 (EudraCT Number)
Record Dates: First submitted 2021-10-28; First posted 2021-11-19 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Neovascular Age-Related Macular Degeneration
Keywords: Wet AMD; neovascular AMD; exudative AMD
MeSH Terms: interventions — Ranibizumab; aflibercept

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Ranibizumab (Experimental): Subjects will have the implant (filled intra-operatively prior to implantation with approximately 20 µL of the 100-mg/mL formulation of ranibizumab [approximately 2-mg dose of ranibizumab]) surgically inserted in the study eye at the Day 1 visit following their randomization visit. Subjects will have their implant refilled with ranibizumab at weeks 36 and 72.
  Interventions: Drug: Ranibizumab; Device: Port Delivery System with ranibizumab (PDS)
- Aflibercept (Active Comparator): Subjects will receive intravitreal injections of aflibercept (2mg) administered in the study eye per treat-and-extend. The decision to extend, maintain, or reduce the interval until next treatment will be per investigator judgment.
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Ranibizumab — Ranibizumab will be administered at a dose of 100 mg/mL delivered via the PDS.
  Arms: Ranibizumab
Drug: Aflibercept — Aflibercept will be administered at a dose of 2 mg in the study eye per treat-and-extend. The decision to extend, maintain, or reduce the interval until next treatment will be per investigator judgment
  Arms: Aflibercept
Device: Port Delivery System with ranibizumab (PDS) — PDS is an investigation intraocular drug delivery device designed to continuously deliver anti-VEGF therapy.
  Arms: Ranibizumab

SUMMARY:
This study will evaluate the effectiveness and safety of a 36-week refill regimen for the Port Delivery System with ranibizumab 100 mg/mL (PDS Q36W) compared with intravitreal injections of aflibercept (2 mg) administered per treat-and-extend (aflibercept T&E) in subjects with neovascular (wet) age-related macular degeneration (nAMD).

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form
2. Age ≥ 50 years, at time of signing Informed Consent Form
3. Ability and willingness to undertake all scheduled visits and assessments
4. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures

   Ocular Inclusion Criteria:
5. Initial diagnosis of nAMD within 9 months prior to the screening visit
6. Previous treatment with at least three anti-VEGF intravitreal injections for nAMD per standard of care within 6 months prior to the screening visit
7. Demonstrated response to prior anti-VEGF intravitreal treatment since diagnosis
8. Availability of historical visual acuity data obtained at or after nAMD diagnosis and prior to the first anti-VEGF treatment for nAMD
9. Availability of historical SD-OCT image data obtained at or after nAMD diagnosis and prior to the first anti-VEGF treatment for nAMD
10. BCVA of 34 letters or better (20/200 or better approximate Snellen equivalent), using ETDRS chart at a starting distance of 4 meters (see the BCVA manual for additional details) at screening and randomization visits
11. With any subtype of nAMD lesions (i.e., type I, type II, type III, or mixed forms per OCT classification, including polypoidal choroidal vasculopathy and retinal angiomatous proliferation)
12. Sufficiently clear ocular media and adequate pupillary dilation to allow for clinical examination and analysis and grading by the central reading center of fundus photography (FP), FA, fundus autofluorescence (FAF) image, and SD-OCT images

Exclusion Criteria:

Prior Ocular Treatment - Study Eye

1. History of vitrectomy surgery, submacular surgery, or other surgical intervention for AMD
2. Prior pars plana vitrectomy surgery
3. Prior treatment with Visudyne® (verteporfin for injection), external-beam radiation therapy, or transpupillary thermotherapy
4. Previous treatment with corticosteroid intravitreal injection
5. Previous intraocular device implantation (not including intraocular lens implants)
6. Previous intraocular surgery (including cataract surgery) within 3 months of randomization
7. Previous laser (any type) used for AMD or diabetic retinopathy treatment
8. History of vitreous hemorrhage
9. History of rhegmatogenous retinal detachment
10. Concurrent conjunctival, Tenon's capsule, and/or scleral condition in the supero temporal quadrant of the eye (e.g., scarring, thinning, mass) that may affect the implantation, subsequent tissue coverage, and refill-exchange procedure of the PDS implant
11. History of glaucoma-filtering surgery, tube shunts, or microinvasive glaucoma surgery
12. History of corneal transplant
13. History of conjunctival surgery in the superotemporal quadrant (including pterygium surgery)

    Prior Ocular Treatment Either Eye:
14. History of a severe allergic reaction or anaphylactic reaction to a biologic agent or known hypersensitivity to any component of the ranibizumab or aflibercept injections, study-related procedure preparations (including fluorescein), dilating drops, or any of the anesthetic and antimicrobial preparations used by a subject during the study
15. Any contraindication to aflibercept as per local label
16. Prior participation in a clinical trial involving any anti-VEGF drugs within 6 months prior to the randomization visit
17. Prior treatment with brolucizumab (at any time prior to the screening visit)
18. Prior treatment with external-beam radiation therapy or brachytherapy

    MNV (CNV) Lesion Characteristics Study Eye:
19. Subretinal hemorrhage that involves the center of the fovea, if the hemorrhage is greater than 0.5-disc area (1.27 mm^2) in size at screening
20. Subfoveal fibrosis or subfoveal atrophy

    MNV (CNV) Lesion Characteristics Either Eye:
21. CNV due to other causes, such as ocular histoplasmosis, trauma, central serous chorio retinopathy, or pathologic myopia
22. CNV masquerading lesions (e.g., cone dystrophy, adult vitelliform dystrophy, pattern dystrophy)

    Concurrent Ocular Conditions Study Eye :
23. Subfoveal and/or juxtafoveal retinal pigment epithelial tear
24. Scleral pathology in the superotemporal quadrant (e.g., scleral thinning or calcification)
25. Conjunctival pathologies (e.g., pterygium, scarring, thinning, fibrosis) in the superotemporal quadrant
26. Any concurrent intraocular condition (e.g., cataract, glaucoma, diabetic retinopathy, epiretinal membrane, amblyopia, or strabismus) that would either require surgical intervention during the study to prevent or treat visual loss that might result from that condition or affect interpretation of study results
27. Active intraocular inflammation (grade trace or above)
28. Rhegmatogenous retinal tears or peripheral retinal breaks on depressed fundus exam that are untreated, or treated within 3 months prior to the randomization visit
29. Aphakia or absence of the posterior capsule Previous violation of the posterior capsule is also an exclusion criterion unless it occurred as a result of yttrium-aluminum garnet (YAG) laser posterior capsulotomy in association with prior, posterior chamber intraocular lens implantation
30. Spherical equivalent of the refractive error demonstrating more than 8 diopters of myopia or evidence of pathologic myopia on depressed fundus exam
31. Preoperative refractive error that exceeds 8 diopters of myopia, for subjects who have undergone prior refractive or cataract surgery in the study eye
32. Spherical equivalent of the refractive error demonstrating more than 5 diopters of hyperopia
33. Preoperative refractive error that exceeds 5 diopters of hyperopia, for subjects who have undergone prior refractive or cataract surgery
34. Uncontrolled ocular hypertension or glaucoma (defined as intraocular pressure [IOP] > 25 mmHg or a cup to disc ratio > 0.8, despite treatment with anti-glaucoma medication) and any such condition the investigator determines may require a glaucoma-filtering surgery during a subject's participation in the study
35. History or presence of severe posterior blepharitis, recurrent chalazia or hordeolum, severe dry eye syndrome, or severe allergic conjunctivitis
36. Ectropion, entropion, ingrowing lashes, or other impairment of the upper or lower eyelid impacting lid functionality needed to protect the ocular surface from exposure
37. Trichiasis
38. Corneal neuropathy
39. Lagophthalmos or incomplete blink
40. Active or history of facial nerve palsy/paresis

    Concurrent Ocular Conditions Non-Study (Fellow) Eye
41. Non-functioning non-study eye, defined as either:

    1. BCVA of hand motion or worse
    2. No physical presence of non-study eye (i.e., monocular)
    3. Legally blind in the subject's relevant jurisdiction

    Concurrent Ocular Conditions Either Eye
42. Any active or history of uveitis (e.g., idiopathic, drug-associated, or autoimmune-associated uveitis)
43. Active or history of keratitis, scleritis, endophthalmitis, or chronic blepharitis
44. Suspected or active ocular or periocular infectious conjunctivitis or endophthalmitis
45. Active or history of Sjogrens syndrome or keratoconjunctivitis sicca
46. Active or history of floppy eyelid syndrome
47. Active or history of chronic eye rubbing
48. Active thyroid eye disease

    Concurrent Systemic Conditions:
49. Inability to comply with study schedule or procedures as described in the study protocol
50. Uncontrolled blood pressure (defined as systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 110 mmHg, while a subject is at rest) If a subject's initial measurement exceeds these values, a second reading should be taken ≥ 30 minutes after the first reading If the subject's blood pressure must be controlled by antihypertensive medication, the subject may become eligible if medication is taken continuously for at least 30 days prior to Day 1
51. Active or history of autoimmune diseases, for example, rheumatoid arthritis, lupus, granulomatosis with polyangiitis (Wegner's)
52. History of stroke within the last 3 months prior to informed consent
53. Atrial fibrillation diagnosed or worsened within the last 3 months prior to informed consent
54. History of myocardial infarction within the last 3 months prior to informed consent
55. History of other disease, metabolic dysfunction (including uncontrolled diabetes), or clinical laboratory finding (after reviewing the results of the screening laboratory results) giving reasonable suspicion of a disease or condition that contraindicates the use of ranibizumab, aflibercept, or placement of the implant and that might affect interpretation of the results of the study or renders the subject at high risk of treatment complications in the opinion of the investigator
56. Confirmed active systemic infection
57. Use of any systemic anti-VEGF agents
58. Chronic use of oral corticosteroids (> 10 mg/day of prednisone or equivalent)
59. Active cancer within 12 months of randomization except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, and prostate cancer with a Gleason score of ≤ 6 and a stable prostate-specific antigen for > 12 months
60. Previous participation in any non-ocular (systemic) disease studies of investigational drugs within 1 month preceding the informed consent (excluding vitamins and minerals)
61. Use of antimitotic or antimetabolite therapy within 30 days or 5 elimination half-lives of the randomization visit
62. Requirement for continuous use of any medications or treatments prohibited in the study
63. Pregnant or breastfeeding, or intending to become pregnant during the treatment period and for at least 3 months after the final intravitreal injection of ranibizumab or aflibercept, or 1 year after the last implant refill-exchange procedure

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12-29 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in BCVA score at week 80 as assessed using the ETDRS visual acuity chart at a starting distance of 4 meters | From baseline up to 80 weeks
  *Depending on the T&E schedule, some subjects in the comparator arm will have a visit at Week 76 and some at Week 78. All subjects in both arms will have a Week 80 visit
Treatment burden as assessed by the treatment frequency up to Week 80 | From baseline up to 80 weeks
  Treatments include injections and refills.

SECONDARY OUTCOMES:
Proportion of subjects with BCVA score of 69 letters (approximate 20/40 Snellen equivalent) or better averaged over Weeks 76 (or 78*) and 80 | Baseline, Week 76, Week 78, Week 80
  *Depending on the T&E schedule, some subjects in the comparator arm will have a visit at Week 76 and some at Week 78. All subjects in both arms will have a Week 80 visit
Proportion of subjects with BCVA score of 38 letters (approximate 20/200 Snellen equivalent) or worse averaged over Weeks 76 (or 78*) and 80 | Baseline, Week 76, Week 78, Week 80
  *Depending on the T&E schedule, some subjects in the comparator arm will have a visit at Week 76 and some at Week 78. All subjects in both arms will have a Week 80 visit
Proportion of subjects who lose < 15, < 10, or < 5 letters in BCVA score from baseline averaged over Weeks 76 (or 78*) and 80 | Baseline, Week 76, Week 78, Week 80
  *Depending on the T&E schedule, some subjects in the comparator arm will have a visit at Week 76 and some at Week 78. All subjects in both arms will have a Week 80 visit
Change from baseline in center point thickness (CPT) at Week 80 | Baseline, Week 80
  *CPT defined as the retinal thickness in the center point of the fovea measured between the internal limiting membrane and the inner third of the retinal pigment epithelium layer, on spectral-domain optical coherence tomography (SD-OCT)
Change from baseline in center subfield thickness (CST), defined as the average thickness of the central 1 mm circle of the ETDRS grid centered on the fovea measured between the internal limiting membrane and the Bruch's membrane, on SD-OCT at Week 80 | Baseline, Week 80
Proportion of subjects randomized to PDS Q36W who do not undergo supplemental treatment with intravitreal ranibizumab 0.5 mg before each refill-exchange procedure | Baseline, Week 80
Incidence and severity of ocular and systemic (non-ocular) adverse events | Baseline, Week 80
Incidence, severity, and duration of adverse events of special interest, including ocular adverse events of special interest | Baseline, Week 80
Incidence, severity, and duration of ocular adverse events of special interest during the postoperative period (≤ 37 days of initial implantation) and follow-up period (> 37 days after implantation surgery) | Baseline, Week 80
Incidence and severity of adverse device effects with PDS Q36W | Baseline, Week 80
Incidence, causality, severity, and duration of anticipated serious adverse device effects with PDS Q36W | Baseline, Week 80

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- Oftalmos, Capital Federal, Argentina
- Denmark (2):
  - Rigshospitalet Glostrup; Afdeling for Øjensygdomme, Glostrup Municipality
  - Sjællands Universitetshospital, Roskilde; Øjenafdelingen, Roskilde
- University Hospital of Larissa; Department of Ophthalmology, Larissa, Greece
- Hong Kong (2):
  - Queen Mary Hospital; Department of Ophthalmology, Hong Kong
  - Hong Kong Eye Hospital; CUHK Eye Centre, Mong Kok
- Hospital de Sao Joao; Servico de Oftalmologia, Porto, Portugal
- Hospital de la Arruzafa. Servicio de Oftalmologia, Córdoba, Spain
- Thailand (2):
  - King Chulalongkorn Memorial Hospital; Ophthalmology Department, Bangkok
  - Maharaj Nakorn ChiangMai Hospital; Ophthalmology Department, Chiang Mai

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on Sharing of Clinical Study Information and how to request access to related clinical study documents, see here (https://www.roche.com/innovation/process/clinical-trials/data-sharing/).